CLINICAL TRIAL: NCT00819754
Title: A Phase I/II Clinical Trial of Combination of Irinotecan, Xeloda and Oxaliplatin (IXO) Regimen With Avastin (Bevacizumab) in Patients With Metastatic Colorectal Cancer
Brief Title: A Phase I/II Study of IXO With Bevacizumab in Patients With Metastatic Colorectal Cancer
Acronym: IXO+A
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Hoffmann-La Roche (Industry); Pfizer (Industry); Sanofi (Industry); Ottawa Regional Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0TT 03-03
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IXO regimen + bevacizumab (Experimental): This is phase I/II safety and efficacy study. There is only one arm of Irinotecan, Xeloda and Oxaliplatin (IXO) regimen with Avastin (bevacizumab)
  Interventions: Drug: IXO regimen + bevacizumab

INTERVENTIONS:
Drug: IXO regimen + bevacizumab — Phase I study - identifies the safety of IXO with bevacizumab and recommended phase II dose
  Phase II study - assesses efficacy and safety of IXO with bevacizumab
  Other Names: irinotecan - Camptosar; capecitabine - Xeloda; Oxaliplatin - Eloxatin; bevacizumab - Avastin

SUMMARY:
Triplets of irinotecan, oxaliplatin and infusional 5-fluorouracil(FU)/leucovorin (LV) are associated with high response rates and long survival as first-line treatment for metastatic colorectal cancer (mCRC). The oral fluoropyrimidine, capecitabine, is better tolerated and shows better response rates than 5-FU/LV in metastatic colorectal cancer. A phase I dose-escalation study established dose limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended phase II doses (RPIID) of irinotecan, oxaliplatin and capecitabine. This phase I /II study is to determine dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), phase II recommended dose (RD) of IXO and bevacizumab combination and safety at the RD in an expanded cohort.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the colon or rectum.
* Advanced and/or metastatic disease, incurable with standard therapy.
* Unresectable advanced and/or metastatic unidimensionally measurable disease (RECIST scale).
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Age: over 18 years.
* Adequate haematological, renal and hepatic functions
* Patient consent must be obtained according to local REB requirements.
* Patients must be accessible for treatment and follow up.

Exclusion Criteria:

* Previous or concurrent malignancies
* Pregnant or lactating women. Women of childbearing potential must have had a negative pregnancy test within 7 days prior to registration.
* Concurrent treatment with other experimental drugs or anticancer therapy.
* Previous chemotherapy for advanced and/or metastatic disease.
* Previous adjuvant therapy with irinotecan or oxaliplatin.
* Previous full dose curative pelvic radiation therapy.
* Patients with documented brain metastases.
* Serious illness or medical condition.
* Gilbert's disease
* Use of enzyme inducing anticonvulsants such as phenytoin, phenobarbital and carbamazepine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-11; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Phase I: Assess the MTD and RD for phase II of IXO and bevacizumab combination given every 3 weeks in 1st line patients with mCRC | 3-week cycle, continuous monitoring of AE
Phase II: Using the RD established in phase I, assess efficacy of the IXO with bevacizumab combination as measured by progression-free survival | 3-week cycle, continuous monitoring of AE

SECONDARY OUTCOMES:
Response rates and duration of response | every 2 cycles - 6 weeks
Overall survival | continuous
Qualitative and quantitative toxicity | continuous

CONTACTS AND LOCATIONS:
Overall Officials: Jean Maroun, MD, Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada